CLINICAL TRIAL: NCT06498453
Title: A Randomized Clinical Trial to Evaluate the Effectiveness of Telerehabilitation With Trak in Patients With Knee or Shoulder Pathology.
Brief Title: Effectiveness of Telerehabilitation With Trak in Knee and Shoulder Pathology: A Randomized Clinical Trial
Acronym: TRAK-TEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trak Health Solutions S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAK-TEST
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Shoulder Injury; Knee Injury
Keywords: Telemedicine; Digital health; Telehealth care
MeSH Terms: conditions — Shoulder Injuries; Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Knee treatment (Experimental): Use of TRAK platform as a treatment metodology on knee patients
  Interventions: Device: Trak-Physio knee condition
- Knee control (Active Comparator): They did not have access to the platform and were instructed to continue with the standard care program through exercise.
  Interventions: Other: Knee conventional rehabilitation program
- Shoulder treatment (Experimental): Use of TRAK platform as a treatment metodology on shoulder patients
  Interventions: Device: Trak-Physio in shoulder condition
- Shoulder control (Active Comparator): They did not have access to the platform and were instructed to continue with the standard care program through exercise.
  Interventions: Other: Shoulder conventional rehabilitation program

INTERVENTIONS:
Device: Trak-Physio knee condition — The exercise protocol designed for knee conditions is carried out through Trak, the digital rehabilitation tool.
  Arms: Knee treatment
Device: Trak-Physio in shoulder condition — The exercise protocol designed for knee conditions is carried out through Trak, the digital rehabilitation tool.
  Arms: Shoulder treatment
Other: Knee conventional rehabilitation program — Exercise protocol with the methodology of conventional clinical practice.
  Arms: Knee control
Other: Shoulder conventional rehabilitation program — Exercise protocol with the methodology of conventional clinical practice.
  Arms: Shoulder control

SUMMARY:
The main objective of this clinical trial is to compare the effectiveness of digital physiotherapy treatment using the Trak telerehabilitation platform and the application of conventional means on two different health conditions (mild or moderate knee osteoarthritis and shoulder tendinopathy)

Participants will undergo telerehabilitation treatment through the TRAK platform for six weeks (treatment group) or follow the instructions and guidelines collected by health personnel for the same time in face-to-face rehabilitation sessions (control group).

DETAILED DESCRIPTION:
The recruitment process for this study is aimed at adults who suffer from musculoskeletal pathologies of the knee (mild or moderate osteoarthritis) or shoulder (tendinopathy).

After the initial screening, individuals who meet the study's predefined inclusion criteria will be invited to participate. Before enrollment, written informed consent will be obtained from all participants, ensuring ethical compliance and respect for individual autonomy.

The study cohort will consist of patients randomly assigned to the experimental group (EG) and the control group (CG) on both knee and shoulder groups. This randomised controlled trial has a parallel design with two groups. Regardless of group assignment, all patients will undergo baseline health assessments, ensuring that their individual needs are met. The satisfaction questionnaire will be deferred until post-intervention for both groups.

Patients will undergo 4 weeks of treatment through the TRAK tool (https://www.trakphysio.com/es/). Patients from the EG will carry out the treatment through the platform at home, and those from the CG will follow an on paper exercise protocol based on the usual (in-person) clinical practice methodology. Both groups will perform exercises in these rehabilitation sessions to improve shoulder mobility.

In phase 1 (3 weeks), all groups will undergo two weeks of in-person treatment based on established drainage technique and TENS application, ensuring the treatment's safety and efficacy. In addition, the patients will begin with in-person (CG) or remote treatment (EG), depending on the case. In the second phase or phase 2 (3 more weeks), patients will perform the exercises at home (EG) or at the medical center (CG).

The results will be evaluated using different scales, such as the DASH scale and the KOOS-PS scale, as well as other secondary scales assessing strength, mobility, pain, and patient satisfaction. These measurements will be collected at the beginning and end of the proposed treatment. These scales will be completed on paper at the beginning and end of the study for both groups, although the daily scales (pain, mobility and strength) will be completed through the platform in the case of the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age.
* Patients with musculoskeletal pathology according to:

Knee: patients between 50 and 70 years old with a knee injury. Among the injuries Considered include mild or moderate osteoarthrosis and knee meniscopathies.

Shoulder: patients with shoulder tendonitis.

* Patients with a tablet, smartphone or laptop who function agilely with the telematic technology necessary for the study.
* Have an email account.
* Understand the purpose of the study.
* Signing of the informed consent.
* Commitment to carry out the prescribed treatments.

Exclusion Criteria:

* Patients with advanced cognitive impairment.
* Patients with tendon tears or ruptures, in patients with shoulder tendinopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Escala DASH | Baseline and six months
  It is used to measure the self-rated upper-extremity disability and symptoms.
Escala KOOS-PS | Baseline and six months
  It evaluates the patient's opinion about their knee and associated problems.

SECONDARY OUTCOMES:
Daniels scale | Baseline and six months
  It is used to measure the patients strength on a specific movement and muscle from 0 to 5, being 0 a total paralysis and a 5 the full joint movement with a resistance.
EVA scale | Baseline and six months
  It is used to measure the level of pain the patient feels.
Trak designed a satisfaction questionnaire | Baseline and six months
  The trak satisfaction questionnaire was provided to patients in Spanish and consists of 12 questions about usability, usefulness and satisfaction as well as a suggestions section at the end.
Limb mobility | Baseline and six months
  It will be measured with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: María A García Velázquez, Principal Investigator — Asunción Klinika
Locations (1):
- Asunción Klinika, Tolosa, Gipuzkoa, Spain

REFERENCES:
- [Background] Anton D, Berges I, Bermudez J, Goni A, Illarramendi A. A Telerehabilitation System for the Selection, Evaluation and Remote Management of Therapies. Sensors (Basel). 2018 May 8;18(5):1459. doi: 10.3390/s18051459. PMID 29738442
- [Background] Chae SH, Kim Y, Lee KS, Park HS. Development and Clinical Evaluation of a Web-Based Upper Limb Home Rehabilitation System Using a Smartwatch and Machine Learning Model for Chronic Stroke Survivors: Prospective Comparative Study. JMIR Mhealth Uhealth. 2020 Jul 9;8(7):e17216. doi: 10.2196/17216. PMID 32480361
- [Background] Cottrell MA, Hill AJ, O'Leary SP, Raymer ME, Russell TG. Service provider perceptions of telerehabilitation as an additional service delivery option within an Australian neurosurgical and orthopaedic physiotherapy screening clinic: A qualitative study. Musculoskelet Sci Pract. 2017 Dec;32:7-16. doi: 10.1016/j.msksp.2017.07.008. Epub 2017 Aug 1. PMID 28787636
- [Background] Cramer SC, Dodakian L, Le V, See J, Augsburger R, McKenzie A, Zhou RJ, Chiu NL, Heckhausen J, Cassidy JM, Scacchi W, Smith MT, Barrett AM, Knutson J, Edwards D, Putrino D, Agrawal K, Ngo K, Roth EJ, Tirschwell DL, Woodbury ML, Zafonte R, Zhao W, Spilker J, Wolf SL, Broderick JP, Janis S; National Institutes of Health StrokeNet Telerehab Investigators. Efficacy of Home-Based Telerehabilitation vs In-Clinic Therapy for Adults After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Sep 1;76(9):1079-1087. doi: 10.1001/jamaneurol.2019.1604. PMID 31233135
- [Background] Hosseiniravandi M, Kahlaee AH, Karim H, Ghamkhar L, Safdari R. Home-based telerehabilitation software systems for remote supervising: a systematic review. Int J Technol Assess Health Care. 2020 Apr;36(2):113-125. doi: 10.1017/S0266462320000021. Epub 2020 Mar 10. PMID 32151291
- [Background] Hung M, Bounsanga J, Voss MW, Saltzman CL. Establishing minimum clinically important difference values for the Patient-Reported Outcomes Measurement Information System Physical Function, hip disability and osteoarthritis outcome score for joint reconstruction, and knee injury and osteoarthritis outcome score for joint reconstruction in orthopaedics. World J Orthop. 2018 Mar 18;9(3):41-49. doi: 10.5312/wjo.v9.i3.41. eCollection 2018 Mar 18. PMID 29564213
- [Background] Monticone M, Baiardi P, Vanti C, Ferrari S, Pillastrini P, Mugnai R, Foti C. Responsiveness of the Oswestry Disability Index and the Roland Morris Disability Questionnaire in Italian subjects with sub-acute and chronic low back pain. Eur Spine J. 2012 Jan;21(1):122-9. doi: 10.1007/s00586-011-1959-3. Epub 2011 Aug 8. PMID 21823035
- [Background] Perruccio AV, Stefan Lohmander L, Canizares M, Tennant A, Hawker GA, Conaghan PG, Roos EM, Jordan JM, Maillefert JF, Dougados M, Davis AM. The development of a short measure of physical function for knee OA KOOS-Physical Function Shortform (KOOS-PS) - an OARSI/OMERACT initiative. Osteoarthritis Cartilage. 2008 May;16(5):542-50. doi: 10.1016/j.joca.2007.12.014. Epub 2008 Feb 21. PMID 18294869
- [Background] Seron P, Oliveros MJ, Gutierrez-Arias R, Fuentes-Aspe R, Torres-Castro RC, Merino-Osorio C, Nahuelhual P, Inostroza J, Jalil Y, Solano R, Marzuca-Nassr GN, Aguilera-Eguia R, Lavados-Romo P, Soto-Rodriguez FJ, Sabelle C, Villarroel-Silva G, Gomolan P, Huaiquilaf S, Sanchez P. Effectiveness of Telerehabilitation in Physical Therapy: A Rapid Overview. Phys Ther. 2021 Jun 1;101(6):pzab053. doi: 10.1093/ptj/pzab053. PMID 33561280
- [Background] van Egmond MA, van der Schaaf M, Vredeveld T, Vollenbroek-Hutten MMR, van Berge Henegouwen MI, Klinkenbijl JHG, Engelbert RHH. Effectiveness of physiotherapy with telerehabilitation in surgical patients: a systematic review and meta-analysis. Physiotherapy. 2018 Sep;104(3):277-298. doi: 10.1016/j.physio.2018.04.004. Epub 2018 Jun 19. PMID 30030037